CLINICAL TRIAL: NCT00074425
Title: Phase II/IIb Safety and Effectiveness Study of the Vaginal Microbicides BufferGel and 0.5% PRO 2000/5 Gel (P) for the Prevention of HIV Infection in Women
Brief Title: BufferGel and PRO 2000/5: Vaginal Gels to Prevent HIV Infection in Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); HIV Prevention Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HPTN 035; 10065 (Registry Identifier: DAIDS ES); NCT00197665 (obsolete NCT alias)
Record Dates: First submitted 2003-12-11; First posted 2003-12-15 (Estimated); Last update posted 2021-11-08 (Actual); Status verified 2013-07

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; Anti-Infective Agents, Local; BufferGel; PRO 2000; Vagina; Risk Factors
MeSH Terms: conditions — HIV Infections | interventions — BufferGel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 1 (Experimental): BufferGel
  Interventions: Drug: BufferGel
- 2 (Experimental): Pro 2000/5 Gel (P)
  Interventions: Drug: PRO 2000/5 Gel
- 3 (Placebo Comparator): Placeo Gel
  Interventions: Drug: Placebo gel
- 4 (No Intervention)

INTERVENTIONS:
Drug: BufferGel — Participants will be given single-use, prefilled applicators of gel and will be instructed to apply one dose of BufferGel intravaginally up to 60 minutes before each vaginal intercourse while in the study.
  Arms: 1
Drug: PRO 2000/5 Gel — Participants will be given single-use, prefilled applicators of gel and will be instructed to apply one dose of PRO 2000/5 Gel intravaginally up to 60 minutes before each vaginal intercourse while in the study.
  Arms: 2
Drug: Placebo gel — Participants will be given single-use, prefilled applicators of gel and will be instructed to apply one dose of PRO 2000/5 Gel intravaginally up to 60 minutes before each vaginal intercourse while in the study.
  Arms: 3

SUMMARY:
The majority of HIV infected people worldwide became infected with the virus through heterosexual contact. BufferGel and PRO 2000 Gel are vaginal gels designed to prevent women from becoming infected with HIV during sexual intercourse with an HIV infected partner. This study will test the safety and effectiveness of these gels.

DETAILED DESCRIPTION:
Accessible, usable, and effective vaginal microbicides could significantly decrease the spread of HIV. Vaginal microbicides could be used with condoms to prevent HIV infection; they could also be used in situations in which an individual is unable to negotiate condom use. Vaginal microbicides are potentially bidirectional, preventing both male-to-female and female-to-male HIV transmission. This study will evaluate the safety and effectiveness of two vaginal microbicides, BufferGel and PRO 2000/5, in preventing the transmission of HIV. The study will also evaluate the effectiveness of these gels in preventing other common sexually transmitted infections (STIs).

BufferGel is a buffering agent designed to maintain normal vaginal acidity in the presence of ejaculate. Studies have shown that HIV is inactivated below a pH of 4 to 5.8. Carbopol 974, the major nonaqueous component of BufferGel, is commonly used as a gelling or tableting agent and has a well-documented safety record. BufferGel has proven safe and well tolerated in Phase I studies. PRO 2000/5 inhibits viral entry into susceptible cells. PRO 2000/5 has also been evaluated in Phase I studies and was found to be safe and well tolerated.

Participants in this study will be randomly assigned to receive one of four interventions: BufferGel, PRO 2000/5, placebo gel, or no gel. All participants will receive HIV risk reduction counseling, condoms, and diagnosis and treatment of sexually transmitted diseases. Participants in the three gel arms will be given single-use, prefilled applicators of gel and will be instructed to apply one dose of the product (BufferGel, PRO 2000/5, or placebo gel) intravaginally up to 60 minutes before each vaginal intercourse while in the study.

Participants will be enrolled for approximately 12 to 30 months, depending on when they enter the study. Participants will have two screening study visits and then monthly visits. Monthly study visits may take place at a clinic, the participant's home, or other community site. Monthly visits will include a medical interview; urine testing, including pregnancy testing; HIV and sexually transmitted infection risk reduction counseling; and distribution of study supplies (condoms and gel-filled applicators). Blood collection will occur at selected monthly visits. Four times a year, participants will be seen in the clinic for a more structured medical interview, pelvic exam, and HIV testing. At one of these visits, participants at particular sites who are willing will be asked to complete a behavioral risk assessment. At some visits vaginal fluid swabs will occur. Participants at non-US study sites will be asked for permission for these swabs to be stored for further testing. Assessment interviews will be both face to face and self-reporting.

ELIGIBILITY:
Note: Per the 12/15/06 amendment, all study participants will now enter the Phase IIb study.

Inclusion Criteria:

* HIV uninfected
* Have had sexual intercourse at least once in the 3 months prior to study entry
* Able to provide adequate contact information to study officials for purposes of follow-up

Exclusion Criteria:

* History of adverse reaction to latex
* Nonmedical injection drug use in the 12 months prior to study entry
* Vaginal intercourse more than an average of two times per day in the 2 weeks prior to study entry
* Plan to become pregnant in the 30 months after study entry
* Plan to travel away from the study site for more than 3 consecutive months in the 30 months after study entry
* Plan to relocate away from the study site in the 30 months after study entry
* Participation in another clinical trial of a vaginal product
* Pregnant within 42 days of study entry
* Have a sexually transmitted disease or other reproductive tract infection diagnosed by study staff
* Abnormal pelvic exam indicating deep epithelial disruption
* Condition that, in the opinion of the investigator, may interfere with the study
* Liver or kidney function abnormality of Grade 3 or higher
* Blood or blood clotting abnormality of Grade 4 or higher

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3101 (Actual)
Dates: Start 2005-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Safety of BufferGel and 0.5% PRO 2000/5 Gel (P), as assessed by deep epithelial disruption, other genital symptoms, or other systemic symptoms | Throughout study
HIV infection as measured by seroconversion | Throughout study

SECONDARY OUTCOMES:
Bacterial vaginosis | Throughout study
Chlamydia infection | Throughout study
Genital ulcer disease | Throughout study
Gonorrhea infection | Throughout study
Herpes simplex virus-2 infection | Throughout study
Pregnancy | Throughout study
Syphilis infection | Throughout study
Trichomoniasis | Throughout study
Acceptability of study product | At Month 3 and study exit
Number of behavioral risk assessment questions not answered in self-reported interviews | Throughout study
Rates of condom use versus gel use | Throughout study
Establishment of a repository of vaginal swab specimens for long-term storage and future research testing on biomarkers of microbicide safety and effectiveness | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Salim Abdool Karim, MBChB, PhD, Study Chair — University of KwaZulu-Natal, Centre for the AIDS Programme of Research in South Africa, Doris Duke Medical Research Institute, Nelson R. Mandela School of Medicine; Irving Hoffman, PA, MPH, Study Chair — School of Medicine, University of North Carolina; Lisa Maslankowski, MD, Study Chair — University of Pennsylvania; Groesbeck Parham, MD, Study Chair — Centre for Infectious Disease Research in Zambia; Nancy Padian, PhD, Study Chair — Department of Obstetrics, Gynecology, and Reproductive Sciences, University of California, San Francisco; AIDS Research Institute; Gita Ramjee, PhD, Study Chair — Medical Research Council, HIV Prevention Research Unit; Taha Taha, MD, Study Chair — Johns Hopkins Bloomberg School of Public Health
Locations (8):
- 3535 Market Street CRS, Philadelphia, Pennsylvania, United States
- Malawi (2):
  - University of North Carolina Lilongwe CRS, Lilongwe, Central Region
  - College of Med. JHU CRS, Blantyre, Southern Region
- South Africa (2):
  - Chatsworth CRS, Chatsworth, KwaZulu-Natal
  - Med. Research Council-Hlabisa, Durban, KwaZulu-Natal
- Kamwala Clinic CRS, Lusaka, Zambia
- Zimbabwe (2):
  - Seke South CRS, Chitungwiza
  - Spilhaus CRS, Harare

REFERENCES:
- [Background] Mayer KH, Peipert J, Fleming T, Fullem A, Moench T, Cu-Uvin S, Bentley M, Chesney M, Rosenberg Z. Safety and tolerability of BufferGel, a novel vaginal microbicide, in women in the United States. Clin Infect Dis. 2001 Feb 1;32(3):476-82. doi: 10.1086/318496. Epub 2001 Jan 26. PMID 11170957
- [Background] van De Wijgert J, Fullem A, Kelly C, Mehendale S, Rugpao S, Kumwenda N, Chirenje Z, Joshi S, Taha T, Padian N, Bollinger R, Nelson K. Phase 1 trial of the topical microbicide BufferGel: safety results from four international sites. J Acquir Immune Defic Syndr. 2001 Jan 1;26(1):21-7. doi: 10.1097/00126334-200101010-00003. PMID 11176265
- [Background] Clarke JG, Peipert JF, Hillier SL, Heber W, Boardman L, Moench TR, Mayer K. Microflora changes with the use of a vaginal microbicide. Sex Transm Dis. 2002 May;29(5):288-93. doi: 10.1097/00007435-200205000-00007. PMID 11984446
- [Background] Tabet SR, Callahan MM, Mauck CK, Gai F, Coletti AS, Profy AT, Moench TR, Soto-Torres LE, Poindexter III AN, Frezieres RG, Walsh TL, Kelly CW, Richardson BA, Van Damme L, Celum CL. Safety and acceptability of penile application of 2 candidate topical microbicides: BufferGel and PRO 2000 Gel: 3 randomized trials in healthy low-risk men and HIV-positive men. J Acquir Immune Defic Syndr. 2003 Aug 1;33(4):476-83. doi: 10.1097/00126334-200308010-00008. PMID 12869836
- [Background] Mayer KH, Karim SA, Kelly C, Maslankowski L, Rees H, Profy AT, Day J, Welch J, Rosenberg Z; HIV Prevention Trials Network (HPTN) 020 Protocol Team. Safety and tolerability of vaginal PRO 2000 gel in sexually active HIV-uninfected and abstinent HIV-infected women. AIDS. 2003 Feb 14;17(3):321-9. doi: 10.1097/00002030-200302140-00005. PMID 12556685
- [Background] D'Cruz OJ, Uckun FM. Clinical development of microbicides for the prevention of HIV infection. Curr Pharm Des. 2004;10(3):315-36. doi: 10.2174/1381612043386374. PMID 14754390
- [Result] MacQueen KM, Namey E, Chilongozi DA, Mtweve SP, Mlingo M, Morar N, Reid C, Ristow A, Sahay S; HPTN 035 Standard of Care Assessment Team. Community perspectives on care options for HIV prevention trial participants. AIDS Care. 2007 Apr;19(4):554-60. doi: 10.1080/09540120601035284. PMID 17453597
- [Result] Minces LR, McGowan I. Advances in the Development of Microbicides for the Prevention of HIV Infection. Curr Infect Dis Rep. 2010 Jan;12(1):56-62. doi: 10.1007/s11908-009-0076-5. PMID 20368766
- [Result] Abdool Karim SS, Richardson BA, Ramjee G, Hoffman IF, Chirenje ZM, Taha T, Kapina M, Maslankowski L, Coletti A, Profy A, Moench TR, Piwowar-Manning E, Masse B, Hillier SL, Soto-Torres L; HIV Prevention Trials Network (HPTN) 035 Study Team. Safety and effectiveness of BufferGel and 0.5% PRO2000 gel for the prevention of HIV infection in women. AIDS. 2011 Apr 24;25(7):957-66. doi: 10.1097/QAD.0b013e32834541d9. PMID 21330907
- [Derived] Guffey MB, Richardson B, Husnik M, Makanani B, Chilongozi D, Yu E, Ramjee G, Mgodi N, Gomez K, Hillier SL, Karim SA; HIV Prevention Trials Network (HPTN) 035 Study Team. HPTN 035 phase II/IIb randomised safety and effectiveness study of the vaginal microbicides BufferGel and 0.5% PRO 2000 for the prevention of sexually transmitted infections in women. Sex Transm Infect. 2014 Aug;90(5):363-9. doi: 10.1136/sextrans-2014-051537. Epub 2014 Jun 4. PMID 24898857
- [Derived] Richardson BA, Kelly C, Ramjee G, Fleming T, Makanani B, Roberts S, Musara P, Mkandawire N, Moench T, Coletti A, Soto-Torres L, Karim SA; HPTN 035 Study Team. Appropriateness of hydroxyethylcellulose gel as a placebo control in vaginal microbicide trials: a comparison of the two control arms of HPTN 035. J Acquir Immune Defic Syndr. 2013 May 1;63(1):120-5. doi: 10.1097/QAI.0b013e31828607c5. PMID 23334506